CLINICAL TRIAL: NCT01747031
Title: Diagnostic Performance of Instantaneous Wave-Free Ratio From Computed Tomography
Brief Title: Determination of Instantaneous Wave-Free Ratio by Computed Tomography
Acronym: iFRCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Ya-Wei Xu, MD FACC, Shanghai 10th People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: Triple | Purpose: Diagnostic
Other Study IDs: NCT20121204
Record Dates: First submitted 2012-12-04; First posted 2012-12-11 (Estimated); Last update posted 2012-12-11 (Estimated); Status verified 2012-12

CONDITIONS: Coronary Artery Disease
Keywords: iFR; FFR; instantaneous wave-free ratio; fractional flow reserve
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single arm study (Experimental): Single arm study.The investigators will conducte computed tomography,angiography and FFR measurement during angiography in this single arm.
  Interventions: Device: PressureWire™ Certus(St. Jude Medical Systems, Sweden)

INTERVENTIONS:
Device: PressureWire™ Certus(St. Jude Medical Systems, Sweden) — Fractional flow reserve measured during cardiac catheterization--A pressure-monitoring guidewire(PressureWire Certus, St. Jude Medical Systems, Uppsala, Sweden) will be advanced past the stenosis.

SUMMARY:
The iFRCT study is a prospective, multicenter study to evaluate the diagnostic performance of iFRCT with the use of ≥64-detector row CT scanners for the detection and exclusion of significant obstructive coronary artery disease, defined by invasive fractiona flow reserve (FFR) as the reference standard.

DETAILED DESCRIPTION:
Noninvasive fractional flow reserve (FFR) computed from CT (FFRCT) is a novel method for determining the physiologic significance of coronary artery disease (CAD), and several clinical trials have revealed that the FFRCT has a good correlation with invasive FFR, also use of noninvasive FFRCT plus Computed Tomography (CT ) among stable patients with suspected or known CAD was associated with improved diagnostic accuracy and discrimination vs CT alone for the diagnosis of hemodynamically significant CAD.

The cornerstone of FFR is the linear relationship between pressure and flow under conditions of constant (and minimized) intracoronary resistance, so is FFRCT. Under such conditions, pressure and flow are assumed to be directly proportional, and a decrease in pressure across a stenosis reflects a decrease in blood flow to the dependent myocardium. However, even after administration of potent pharmacologic agents such as adenosine, intracoronary resistance is not static, but instead fluctuates in a phasic pattern throughout the cardiac cycle. In addition, for patients who are allergic to pharmacologic agents or with sever lesions which response little to pharmacologic agents, the measurement of FFR is challenging and the lesion are always underestimated. The ADVISE trial revealed that intracoronary resistance is naturally constant and minimized during the wave-free period. The instantaneous wave-free ratio calculated over this period produces a drug-free index of stenosis severity comparable to FFR. But whether iFR calculated from Computed Tomography(iFRCT) is comparable to FFRCT or FFR, and its diagnostic performance remains unknown. Thus the investigators conduct this trial to assess the diagnostic performance of Instantaneous Wave-Free Ratio for diagnosis of hemodynamically significant coronary stenosis.

Instantaneous Wave-Free Ratio calculated from reconstructed heart model.Wave-intensity analysis identified a wave-free period in which intracoronary resistance at rest is similar in variability and magnitude.The investigators define the resting distal-to-proximal pressure ratio during this period as the instantaneous wave-free ratio (iFR).

ELIGIBILITY:
Inclusion Criteria:

* Coronary computed tomographic angiography(CCTA) with over 50 percent stenosis in a major coronary artery over 2mm diameter
* Undergoing clinically indicated invasive coronary angiography with FFR

Exclusion Criteria:

* A history of CABG surgery
* Prior percutaneous coronary intervention with suspected instent restenosis
* Suspicion of or recent acute coronary syndrome
* Complex congenital heart disease
* Prior pacemaker or defibrillator
* Prosthetic heart valve
* Significant arrhythmia
* heart rate >100 beats/min
* systolic blood pressure≤90 mmHg
* contraindication to beta blockers, nitroglycerin or adenosine
* Serum creatinine level greater than 1.5 mg per dL
* Allergy to iodinated contrast
* Pregnant state
* Body mass index greater than 35
* Evidence of active clinical instability or lifethreatening disease
* Canadian Cardiovascular Society class IV angina
* nonevaluable CCTA as determined by the CCTA core laboratory
* Inability to adhere to study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-12; Primary Completion 2014-06 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Accuracy of iFRCT | 1 day
  Diagnostic accuracy[Sensitivity, specificity, positive predictive value (PPV) and negative predictive value (NPV)]* of CCTA plus iFRCT(instantaneous wave-free ratio calculated in reconstructed heart model) or iFRCT alone to determine presence or absence of at least one hemodynamically (HD)-significant coronary artery stenosis at the subject level using binary outcomes when compared to FFR as the reference standard.*Sensitivity measures the proportion of actual positives which are correctly identified. Specificity measures the proportion of negatives which are correctly identified;PPV, or precision rate is the proportion of positive test results that are true positives (such as correct diagnoses);NPV is defined as the proportion of subjects with a negative test result who are correctly diagnosed.

SECONDARY OUTCOMES:
Diagnostic accuracy of iFRCT at the subject level | 1 day
  Sensitivity, specificity, positive predictive value (PPV) and negative predictive value (NPV) of CCTA plus iFRCT or iFRCT alone at the subject level using binary outcomes when compared to FFR as the reference standard.
Diagnostic accuracy of iFRCT at the vessel level | 1 day
  Sensitivity, specificity, PPV and NPV of CCTA plus iFRCT or iFRCT alone for the presence or absence of HD-significant coronary artery stenosis at the vessel level using binary outcomes when compared to FFR as the reference standard.
FFR Numerical Correlation | 1 day
  Per-vessel correlation of the iFRCT numerical value alone with the FFR numerical value measured during cardiac catheterization.
FFRCT Numerical Correlation | 1 day
  Per-vessel correlation of the iFRCT numerical value alone with the FFRCT numerical value calculated from the computed tomography.
Predicted Post-PCI FFR Measurement | 1 day
  Diagnostic accuracy of predicted post-percutaneous intervention (PCI) iFRCT alone to determine success or failure of PCI* using binary outcomes when compared to post-PCI FFR at the subject and vessel level using PCI as the reference standard.*PCI success will be defined as post-PCI FFR>0.80, while PCI failure will be defined as post-PCI FFR≤0.80 during adenosine-mediated hyperemia.

CONTACTS AND LOCATIONS:
Overall Officials: Ya-Wei Xu, MD, FACC, Principal Investigator — Department of Cardiology, Shanghai Tenth People's Hospital, Tongji University School of Medicine
Locations (1):
- Department of Cardiology, Shanghai Tenth People's Hospital, Shanghai, China

REFERENCES:
- [Background] Sen S, Escaned J, Malik IS, Mikhail GW, Foale RA, Mila R, Tarkin J, Petraco R, Broyd C, Jabbour R, Sethi A, Baker CS, Bellamy M, Al-Bustami M, Hackett D, Khan M, Lefroy D, Parker KH, Hughes AD, Francis DP, Di Mario C, Mayet J, Davies JE. Development and validation of a new adenosine-independent index of stenosis severity from coronary wave-intensity analysis: results of the ADVISE (ADenosine Vasodilator Independent Stenosis Evaluation) study. J Am Coll Cardiol. 2012 Apr 10;59(15):1392-402. doi: 10.1016/j.jacc.2011.11.003. Epub 2011 Dec 7. PMID 22154731